CLINICAL TRIAL: NCT05957302
Title: Comparing the Hemodynamic Effects of Bolus of Ketamine and Fentanyl in Patients With Septic Shock: a Randomized Controlled Trial
Brief Title: Hemodynamic Effects of Bolus of Ketamine Versus Fentanyl in Patients With Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MS-47-2023
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Ketamine; Fentanyl; Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Ketamine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine group (Active Comparator): bolus of sedation for resuming sedation after sedation vacation
  Interventions: Drug: Ketamine
- Fentanyl group (Active Comparator): bolus of sedation for resuming sedation after sedation vacation
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Ketamine — 100 mg of ketamine diluted in 10 mL saline (10 mg /mL) and patient will receive 0.1 mL/kg
  Arms: Ketamine group
Drug: Fentanyl — 100 mcg of fentanyl diluted in 10 mL saline (10 mcg /mL) and patient will receive 0.1 mL/kg
  Arms: Fentanyl group

SUMMARY:
Ketamine is a commonly used drug for sedation and induction of anesthesia in patients with shock and/or cardiac dysfunction. Ketamine is characterized by its cardiovascular stimulatory effect due to increase release of endogenous catecholamines. On the other hand, laboratory data on the isolated human myofibers suggest that ketamine had a direct myocardial depressive effect; accordingly, many experts believe that ketamine might have a negative hemodynamic effect in catecholamine depleted patients such as critically ill patients. In critically ill patients, there are contradicting results for the effect of ketamine on the hemodynamic profile and there is paucity of clinical data about the effect of ketamine on cardiac contractility and cardiac output (CO). Cardiac output is the primary determinant of global oxygen delivery to organs and maintaining stable CO in critically ill patients is at most importance to avoid further organ damage in such patients.

Therefore, this study is designed to evaluate the effect a single bolus of ketamine on CO in patients with septic shock in comparison to fentanyl bolus.

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria will receive the study drug according to the randomization, if a bolus of sedation is required for resuming sedation after sedation vacation. All patients will be monitored by 5-lead electrocardiogram, pulse oximetry, and noninvasive blood pressure.

Hypotension defined as mean arterial pressure < 65 mmHg and will be managed by increasing the norepinephrine infusion rate by 20%.

Bedside echocardiography will be used to measure the cardiac output by an experienced physician who is not aware of the nature of the study drug. The left ventricular outflow diameter (LVOT) will be measured in the parasternal long-axis view. Then velocity time integral (VTI) will be measured from the apical five-chamber view. The average of three VTI readings will be calculated.

The cardiac output will be calculated by the equation:

CO = π X (LVOT diameter/2) X VTI X heart rate Delta CO% will be calculated as percentage of change at each time point in relation to the baseline measurement the CO, heart rate, mean blood pressure will be measured before drug administration and at 3, 6, 10 and 15 min after drug administration

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) patients.
* With septic shock on vasopressor therapy
* Mechanically ventilated
* Need for sedation

Exclusion Criteria:

* Hemodynamic instability (MAP <65 mmHg) despite appropriate volume replacement and vasopressor therapy
* Noradrenaline infusion rate <0.05 mcg/kg/min
* Poor cardiac window on the ultrasound.
* Known allergy to study drugs
* Neurocritical patients with signs of increased intracranial tension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
6-minutes Delta CO% | at 6 minutes after drug administration
  percentage of change at 6 min after drug administration in relation to the baseline measurement

SECONDARY OUTCOMES:
Delta CO% | 3, 6, 10 and 15 minutes after drug administration
  percentage of change at each time point after drug administration in relation to the baseline measurement
heart rate | 3, 6, 10 and 15 minutes after drug administration
  beat per minute
mean blood pressure | 3, 6, 10 and 15 minutes after drug administration
  mmHg
norepinephrine dose | 3, 6, 10 and 15 minutes after drug administration
  mcg/kg/min

CONTACTS AND LOCATIONS:
Overall Officials: ahmed hasanin, MD, Principal Investigator — Cairo University Kasr Alainy Faculty of Medicine
Locations (1):
- Ahmed Mohamed Hasanin, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The datasets used during the current study will be available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Mostafa M, Hasanin A, Reda B, Elsayad M, Zayed M, Abdelfatah ME. Comparing the hemodynamic effects of ketamine versus fentanyl bolus in patients with septic shock: a randomized controlled trial. J Anesth. 2024 Dec;38(6):756-764. doi: 10.1007/s00540-024-03383-9. Epub 2024 Aug 18. PMID 39154316